CLINICAL TRIAL: NCT03820518
Title: Comparing the Effectiveness of High or Low Dose of Active Vitamin D Combined With Neutral Phosphate in Children With X-linked Hypophosphatemia
Brief Title: Using Different Doses of Active Vitamin D Combined With Neutral Phosphate in Children With X-linked Hypophosphatemia
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JS-1824
Record Dates: First submitted 2019-01-25; First posted 2019-01-29 (Actual); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: X-linked Hypophosphatemia
MeSH Terms: conditions — Familial Hypophosphatemic Rickets | interventions — Calcitriol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-dose (Experimental): Receiving 60 ng/kg/day of calcitriol and 30 mg/kg/day of elemental phosphorus.
  Interventions: Drug: Calcitriol
- Low-dose (Experimental): Receiving 20 ng/kg/day of calcitriol and 30 mg/kg/day of elemental phosphorus.
  Interventions: Drug: Calcitriol

INTERVENTIONS:
Drug: Calcitriol
  Other Names: Elementary phosphorus

SUMMARY:
X-linked hypophosphatemia (XLH) is the most common form of heritable rickets. Current treatments include active vitamin D metabolites (e.g. calcitriol) and phosphate salts. There is no consistent weight-based dosing of calcitriol and phosphate now. The primary objective of this study is to establish the efficacy of different dose of calcitriol combined with neutral phosphate in children with XLH.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 1-12 years, inclusive
* Diagnosis of XLH by clinical features: serum phosphorus level < 2.5 mg/dl; ALP?; RSS total score ≥2; bowed legs; short stature; family history with appropriate X-linked inheritance
* Meet at least one of the following: confirmed Phosphate regulating gene with homology to endopeptidases located on the X chromosome (PHEX) mutation in the participant, or serum FGF23 level >30 pg/ml (Kainos assay)
* Willing to participate the study, and provide an informed consent
* Able to complete all aspects of study and adhere to the visit schedule

Exclusion Criteria:

* Use of growth hormone within 12 months before first visit
* Height >50 percentile for age and sex specific data
* Presence of nephrocalcinosis or nephrolithiasis
* Serum intact parathyroid hormone level>170 pg/ml
* Plan to receive orthopaedic surgery in 12 months
* Poor compliance
* Use of gonadotropin-releasing hormone therapy right now
* Use of aluminium hydroxide, steroid, acetazolamide or thiazide drugs within 7 days before first visit
* Not be fit to participant in the study, by the judgement of investigators

Ages: 1 Year to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline to Post-treatment in Severity of Rickets as Measured by Rickets Severity Score (RSS) Total Score | Baseline, Month 12, 24
  RSS range from 0 to 10, and higher RSS represent severer rickets. It is consisted of score of worst wrist (0-4) and worst knee (0-6).
  WRIST-score both radius and ulna separately-2 bones × 2 points = 4 points possible KNEE-score both femur and tibia separately Multiply the grade in A by the multiplier in B for each bone, then add femur and tibia scores together A: Grade
  1 2 3 B: Multiplier Portion of growth plate affected 0.5 ≤ 1 condyle or plateau
  1. 2 condyles or plateaus
  2. bones × 1 point × 3 points = 6 points possible Total: 10 points possible Reference:Thacher, T. Radiographic scoring method for the assessment of the severity of nutritional rickets[J]. Journal of Tropical Pediatrics, 2000, 46(3):132-139.

SECONDARY OUTCOMES:
Changes From Baseline to Post-treatment in Severity of Rickets as Measured by RSS Wrist and Knee Score | Baseline, Month 12, 24
  RSS range from 0 to 10, and higher RSS represent severer rickets. It is consisted of score of worst wrist (0-4) and worst knee (0-6).
  WRIST-score both radius and ulna separately-2 bones × 2 points = 4 points possible KNEE-score both femur and tibia separately Multiply the grade in A by the multiplier in B for each bone, then add femur and tibia scores together A: Grade
  1 2 3 B: Multiplier Portion of growth plate affected 0.5 ≤ 1 condyle or plateau
  1. 2 condyles or plateaus
  2. bones × 1 point × 3 points = 6 points possible Total: 10 points possible Reference:Thacher, T. Radiographic scoring method for the assessment of the severity of nutritional rickets[J]. Journal of Tropical Pediatrics, 2000, 46(3):132-139.
Changes From Baseline to Post-treatment in Growth Velocity | Baseline, Month 12, 24
  Changes From Baseline to Post-treatment in Severity of Rickets as Measured by RSS Wrist and Knee Score
Changes From Baseline to Post-treatment in Serum Total Alkaline Phosphatase (TALP) Levels | Baseline, Month 3, 6, 12, 18, 24
  Changes From Baseline to Post-treatment in serum ALP
Changes From Baseline to Post-treatment in serum Carboxy-terminal Collagen Crosslinks (CTX) Levels | Baseline, Month 3, 6, 12, 18, 24
  Changes From Baseline to Post-treatment in serum CTX
Changes From Baseline to Post-treatment in Serum Phosphorus Levels | Baseline, Month 3, 6, 12, 18, 24
  Changes From Baseline to Post-treatment in Serum Phosphorus Levels
Changes From Baseline to Post-treatment in Severity of Dental Abscess | Baseline, Month 3, 6, 12, 18, 24
  The frequency and number of dental abscess will be collected by self-report and examed by investigators
Changes From Baseline to Post-treatment in Severity of Bone Pain as Measured by Visual Analog Pain Scales | Baseline, Month 3, 6, 12, 18, 24
  Visual Analog Pain Scales (VAS) range from 0-10, and higher score represents severer pain
Changes From Baseline to Post-treatment in Severity of Leg Deformities | Baseline, Month 3, 6, 12, 18, 24
  The longest distance between two sides of thighs, knees, shanks and ankles are measured to evaluate the severity of leg deformities.
Changes From Baseline to Post-treatment in Serum Osteocalcin Levels | Baseline, Month 3, 6, 12, 18, 24
  Changes From Baseline to Post-treatment in Serum Osteocalcin Levels
Changes From Baseline to Post-treatment in Height | Baseline, Month 3, 6, 12, 18, 24
  Changes From Baseline to Post-treatment in Height
Changes From Baseline to Post-treatment in Quality of Life as Measured by Patient-reported Outcomes Measurement Information System | Baseline, Month 3, 6, 12, 18, 24
  Changes From Baseline to Post-treatment in Quality of Life as Measured by Patient-reported Outcomes Measurement Information System

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Endocrinology, Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No